CLINICAL TRIAL: NCT01076062
Title: Elective Induction of Nulliparous Labor: A Randomized Clinical Trial
Brief Title: Elective Induction of Nulliparous Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sandra Smith, Maternal Fetal Medicine Fellow, Madigan Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210013
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy
Keywords: Pregnancy Maintenance; Labor, Induced; spontaneous labor; cesarean delivery
MeSH Terms: interventions — Labor, Induced; Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expectant management (EM) arm (No Intervention): Standard of care: routine clinic appointments until they deliver, fetal heart rate and contraction monitoring during their 41st week if not delivered. Also if they have not gone into labor the subjects will be scheduled for an induction by 42 weeks.
- Induction of Labor (IOL) arm (Experimental): Elective induction of labor at 39 weeks.
  Interventions: Procedure: Induction of Labor

INTERVENTIONS:
Procedure: Induction of Labor — If cervical foley bulb placement is possible, the foley bulb will remain in place until either spontaneously removed or after 12 hrs, whichever is earlier. If placement is not possible, cervical ripening with misoprostol 25 micrograms (mcg) per vagina every 4 hrs (max of 4 total doses) will be initiated. Cervical examination will occur every 4 hr. Repeat doses of misoprostol will be given only if foley bulb placement is not possible and/or if palpably firm uterine contractions are less than 6 in 10 min in consecutive 10 min intervals. Once placement of a cervical foley bulb can be performed, oxytocin administration will begin at 2 mIU/min and increasing by 2 mIU/min every 20 min to ensure adequate contractions (maximum oxytocin infusion rate 36 mIU/min). Adequate contractions will be defined as 7 contractions in 15 min in consecutive 15 min intervals that palpate moderate to firm. Oxytocin infusion will begin not earlier than 4 hrs after the last misoprostol dose (if given).
  Other Names: misoprostol; oxytocin
  Arms: Induction of Labor (IOL) arm

SUMMARY:
Primary outcome: to evaluate the effect of elective induction of labor (IOL), at 39 weeks gestation, on cesarean delivery rates in nulliparous women compared to expectant management (EM).

Secondary outcomes: to evaluate differences in the mean number of clinic visits/antepartum tests avoided with IOL, to compare the differences in utilization of inpatient resources (mean duration of inpatient stay, mean duration of labor), and to evaluate the effect of IOL on the risk of urinary/anal incontinence and sexual dysfunction as analyzed using previously validated measurements. We will evaluate differences in the rate of cervical change once active labor is diagnosed, and the time from completion of active labor, defined as complete dilation and complete effacement, to the delivery of fetus (definition of second stage of active labor). Furthermore, other secondary outcomes to be evaluated include comparisons between IOL and EM in regards to the occurence of chorioamnionitis, stillbirth, operative vaginal delivery, and meconium stained amniotic fluid. An evaluation of the predictive value of cervical length and Bishop score for vaginal delivery will also be examined.

DETAILED DESCRIPTION:
A research nurse will screen patients at the 38 week visit through chart review and potential candidates will be identified. One of the study investigators or research nurse will interface with the patient at the 38 week visit and written informed consent will be obtained after the study protocol is explained and eligibility determined. Since eligibility determination cannot be made without performing a digital cervical examination, the patient will be offered a cervix exam with Bishop score determination. If the Bishop score meets inclusion criteria, the patient will be offered participation in the study. Women who consent to the study will be randomized using a computer-generated list by means of sequentially numbered, opaque, sealed envelopes which reveal the allocation of the subject to either induction or expectant management. All subjects will then receive the following evaluation: transvaginal cervical length measurement, and completion of a standard urinary/rectal incontinence/sexual function questionnaire. Patients randomized to induction will be scheduled not earlier than 39 weeks gestation and in coordination with the labor and delivery physician and nursing leadership. The method of induction will be dependant on whether or not a cervical foley bulb can be placed at the time of admission for induction of labor. If cervical foley bulb placement is possible, the foley bulb will remain in place until either spontaneously removed or after 12 hours, whichever is earlier. If placement is not possible, cervical ripening with misoprostol 25 mcg per vagina every 4 hours (maximum of 4 total doses) will be initiated. Cervical examination will occur every 4 hours (coincident with vaginal misoprostol placement). Repeat doses of misoprostol will be given only if foley bulb placement is not possible and/or if palpably firm uterine contractions are less than 6 in 10 minutes in consecutive 10 minute intervals. Once placement of a cervical foley bulb can be performed this will be accomplished and initiation of oxytocin administration will begin at 2 mIU/minute and increasing by 2 mIU/minute every 20 minutes to ensure adequate contractions (maximum oxytocin infusion rate 36 mIU/minute). Adequate contractions will be defined as 7 contractions in 15 minutes in consecutive 15 minute intervals that palpate moderate to firm. Oxytocin infusion will begin not earlier than 4 hours after the last misoprostol dose (if given). Subjects expectantly managed (EM) will be scheduled for routine follow-up appointments and delivered for obstetric indications but not later than 42 weeks gestation.

A routine 6-8 week immediate postpartum and 1 year follow-up examinations will be scheduled for all subjects following delivery. In addition to the routine examinations, all subject evaluations during these visits will include completion of a standard urinary/rectal incontinence/sexual function.

Study data will be entered into a password protected Excel file on a DoD government computer accessible only to study investigators and a clinical research nurse. Withdrawal from the study will be voluntary and results will be analyzed on an intent-to-treat basis.

Data analysis will focus on the primary outcome: to evaluate the effect of elective induction of labor, at 39 weeks gestation, on cesarean delivery rates in nulliparous women compared to expectant (typical) management. Also evaluation of secondary outcomes will include determination of the predictive value of cervical length and Bishop score for successful vaginal delivery; the risk of urinary/anal incontinence and sexual dysfunction with labor induction compared to spontaneous labor; number of clinic visits/antepartum tests avoided with elective induction compared with potential increased utilization of inpatient resources; evaluation of the labor curve with induction compared to spontaneous labor. Other secondary outcomes to be evaluated include comparisons between IOL and EM in regards to the rate of chorioamnionitis, rate of stillbirth, rate of operative vaginal delivery, and rate of meconium stained amniotic fluid. Students t-test will be used to compare continuous variables and the Chi-square test will be used to compare proportions between the groups. Analysis is by intent-to-treat with a p-value of less than 0.05 considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous patients evaluated at 38 weeks gestation without contraindication for induction of labor, and
* Patients who meet dating criteria as outlined above, and
* Patients who have a Bishop score of ≤ 5.

Exclusion Criteria:

* Contraindication to induction of labor,
* Scheduled induction of labor for medical indications, and/or
* Failure to meet dating criteria above, Bishop score of > 5.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2009-10-27 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Cesarean Birth Rate | 39 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel R Miller, MD, Principal Investigator — Madigan Army Medical Center; Peter Nielsen, MD, Study Director — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Middleton P, Shepherd E, Morris J, Crowther CA, Gomersall JC. Induction of labour at or beyond 37 weeks' gestation. Cochrane Database Syst Rev. 2020 Jul 15;7(7):CD004945. doi: 10.1002/14651858.CD004945.pub5. PMID 32666584
- [Derived] Miller NR, Cypher RL, Foglia LM, Pates JA, Nielsen PE. Elective Induction of Labor Compared With Expectant Management of Nulliparous Women at 39 Weeks of Gestation: A Randomized Controlled Trial. Obstet Gynecol. 2015 Dec;126(6):1258-1264. doi: 10.1097/AOG.0000000000001154. PMID 26551184